CLINICAL TRIAL: NCT06126237
Title: A Phase I/II, Multiple Center, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of CM313 in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of CM313 in Subjects With Relapsed or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM313-040101
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM313 (Experimental): CM313 injection, subcutaneous
  Interventions: Biological: CM313 injection
- CM313 + concomitant medication (Experimental): CM313 injection, subcutaneous
  Interventions: Biological: CM313 injection

INTERVENTIONS:
Biological: CM313 injection — CM313, subcutaneous injection

SUMMARY:
This is a multi-center, open-label, Phase 1/2 study to evaluate the safety, tolerability, Pharmacokinetics, pharmacodynamics and Preliminary Efficacy of CM313 in Subjects with Relapsed or Refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age ≥ 18 years.
* Subjects diagnosed with multiple myeloma.
* Subjects with measurable lesions.
* Women of childbearing potential with negative pregnancy testing.
* Subjects voluntarily signed the Informed Consent Form and were able to comply with the provisions of this protocol.

Exclusion Criteria:

* Previous treatment with any anti-CD38 therapy.
* Vaccinated with live, attenuated vaccine within 4 weeks prior to the first dose.
* Positive for human immunodeficiency virus (HIV) antibodies.
* Syphilis antibody positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-28 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse event | up to 18 months
  Incidence, severity, and outcome of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)